CLINICAL TRIAL: NCT04149457
Title: Improving Neurological Health in Aging Via Neuroplasticity-based Computerized Exercise (INHANCE)
Brief Title: Improving Neurological Health in Aging Via Neuroplasticity-based Computerized Exercise
Acronym: INHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-0903-19
Record Dates: First submitted 2019-10-28; First posted 2019-11-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 70 treatment sessions, up to 7 sessions per week, 30 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training requiring a total maximum of 70 treatment sessions, up to 7 sessions per week, 30 minutes per session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Thirty minutes of training on computerized exercises that targets visual processing speed, memory, attention and alertness.
  Arms: Experimental Treatment
Other: Commercially available computerized training — Thirty minutes of training on computerized, casual video games.
  Arms: Active Comparator

SUMMARY:
This study is a validation study to evaluate efficacy of a neuroplasticity-based, computerized cognitive training program INHANCE (Improving Neurological Health in Aging via Neuroplasticity-based Computerized Exercise) to improve neurological and neuropsychological health in older adults.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the impact of a targeted speed and alertness training program (INHANCE) to improve cognition in healthy older adults, as evidenced by standard measures of cognition, and positive improvements in the neuromodulatory cholinergic system as measured via positron-emission tomography (PET).

The investigators will employ a double-blind, parallel-arm, placebo-controlled, randomized clinical trial design comprised of a treatment group using INHANCE, a computerized program that trains speed of processing and attention, compared to an active control group using computer games in 92 healthy older adults.

Approximately 108 participants will be consented to ensure the successful completion of 92 participants (post 20% attrition). Participants will then complete the Screening (V0) assessments to determine eligibility. Following inclusion, participants will complete the Baseline (V1) assessments, PET imaging and structural MRI scan; participants will then be randomized into either the INHANCE training or Computer Games, and will engage in approximately 35 hours of program use for the 10-week intervention period. Approximately halfway through the intervention period (~5 weeks), participants will complete Interim (V2) assessments to be compared to the Post-Intervention assessments. Following the 10-week intervention, participants will complete a Post-Intervention (V3) assessment and PET imaging to evaluate changes in cognitive function. Participants will then stop using their assigned program for 3 months and return for a Follow-up (V4) end-of-study assessment to evaluate the endurance of changes in cognitive function in the absence of further program use.

The protocol will be conducted in accordance with the protocol submitted to and approved by the National Institute on Health (NIH), and subject to Institutional Review Board review and approval prior to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Potential participant must be 65+ years old at the time of study screening.
* Potential participant should achieve a score of ≥ 23 on the Montreal Cognitive Assessment (MoCA).
* Potential participant must be likely able to compete all primary outcome measures in the judgment of the consenting study staff person.
* Potential participant must demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in this research study.
* Potential participant must have the visual, auditory, and motors capacity to use the computerized intervention in the judgment of the consenting study staff person.
* Potential participant must already have, be willing to obtain, or be willing to travel to locations with WiFi connectivity to complete intervention activities.
* Potential participant must be able to communicate in either English or French.

Exclusion Criteria:

* Potential participant should not have an existing diagnosis of major or minor neurocognitive disorder at screening.
* Potential participants with active suicidal ideation with specific plan and intent or suicide-related behaviors within 2 months of consent as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Potential participant should not have a Geriatric Depression Scale (GDS) score of >10.
* Potential participant should not have been treated within 5 years of the date of consent with a computer-based cognitive training program manufactured by Posit Science.
* Potential participant should not be participating in a concurrent clinical trial (involving an investigational pharmaceutical, behavioral treatment, medical device or other) that, in the judgment of the Site Principal Investigator, could affect the outcome of this study.
* Potential participant may not be pregnant and should not have claustrophobia or implantation with any medical devices above the waist that may concentrate radio frequency fields, or have other medical issues that may frustrate participation in MRI imaging procedures.
* Potential participant should not have medical illnesses deemed to interfere with participation in study activities and/or unstable and/or untreated conditions that may affect cognition, including substance abuse/dependence disorders, drugs that interfere with cholinergic function, ongoing chemotherapy or other cancer treatment.
* Potential participant who shows signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs) will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Change in FEOVB uptake through PET Imaging | At 3 months (post-intervention)
  18F-fluoroethoxybenzovesamicol (FEOBV) uptake as measured through Positron Emission Tomography (PET) ligand imaging.

OTHER OUTCOMES:
Change in EXAMINER Executive Composite Score | At 3 months (post-intervention) and at 6 months (follow-up)
  The EXAMINER is a computer based battery of executive function tests which yields a total or 'composite' score to represent global executive functioning. Executive composite scores can range from -3.0 to 3.0 with higher scores corresponding to better executive functioning, and negative scores indicating impairment.
Change in Useful Field of View (UFOV) Score | At 3 months (post-intervention) and at 6 months (follow-up)
  This is a computerized assessment that serves as a positive control for task learning. A single exposure duration (in milliseconds) required for users to achieve approximately 80% criterion accuracy in identification of central and peripheral targets. The score range is 10ms - 5000ms (lower scores indicate better performance).
Change in Tonic and Phasic Alertness (TAPAT) Score | At 0 months (pre-intervention), at 3 months (post-intervention) and at 6 months (follow-up)
  This is a computerized assessment that serves as a positive control for task learning. A single target frequency required for users to achieve at least 80% accuracy in target and foil identification for a pre-specified target image presented among similar foil images. The score range is 1-7 corresponding to 40%, 35%, 30%, 25%, 20%, 15%, and 10% target frequencies (higher scores indicate better performance).
Change in Heart Rate Variability | At 3 months (post-intervention) and at 6 months (follow-up)
  Heart rate variability will be measured to determine acetylcholinergic function over time.
Change in Pupillometry | At 3 months (post-intervention) and at 6 months (follow-up)
  Pupil dilation will be measured to determine acetylcholinergic function over time.
Stricture and Resting through MRI Imaging | At 3 months (post-intervention)
  Stricture and resting will be observed through MRI Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation; Mouna Attarha, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attarha M, de Figueiredo Pelegrino AC, Toussaint PJ, Grant SJ, Van Vleet T, de Villers-Sidani E. Improving Neurological Health in Aging Via Neuroplasticity-Based Computerized Exercise: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Aug 8;13:e59705. doi: 10.2196/59705. PMID 39116435
- [Derived] Attarha M, de Figueiredo Pelegrino A, Ouellet L, Toussaint PJ, Grant SJ, Van Vleet T, de Villers-Sidani E. Effects of Computerized Cognitive Training on Vesicular Acetylcholine Transporter Levels using [18F]Fluoroethoxybenzovesamicol Positron Emission Tomography in Healthy Older Adults: Results from the Improving Neurological Health in Aging via Neuroplasticity-based Computerized Exercise (INHANCE) Randomized Clinical Trial. JMIR Serious Games. 2025 Oct 13;13:e75161. doi: 10.2196/75161. PMID 41084791
- See also: Two years after trial completion (on May 31, 2026), the INHANCE dataset will be made available to verified academic and industry researchers. Investigators can conduct both confirmatory and exploratory analyses using LORIS. — https://inhance.loris.ca/